CLINICAL TRIAL: NCT06625047
Title: Neuro-Oncology Anywhere 242: Pilot Study Evaluating Telehealth and In-Person Assessments in Patients With Glioma Receiving Oral Chemotherapy
Brief Title: Comparing Telehealth and In-person Assessments in Glioma Patients Receiving Oral Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NOA242; NCI-2024-07700 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NOA242 (Other: Mayo Clinic Neuro-Oncology); 24-007538 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Astrocytoma, IDH-Mutant; Glioblastoma; Glioma; Oligodendroglioma, IDH-Mutant and 1p/19q-Codeleted
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma; Oligodendroglioma | interventions — Restraint, Physical; Outcome Assessment, Health Care; Observational Studies as Topic; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (temozolomide, telehealth, in-person) (Experimental): Patients receive temozolomide PO QD on days 1-5 of each cycle. Cycles repeat every 28 days for up to 6 cycles while on study in the absence of disease progression or unacceptable toxicity. Patients complete alternating telehealth assessment visits and in-person assessment visits after each cycle of treatment.
  Interventions: Behavioral: Assessment; Other: Questionnaire Administration; Other: Telemedicine Visit; Drug: Temozolomide

INTERVENTIONS:
Behavioral: Assessment — Complete in-person assessment visits
  Other Names: Assess; Study Assessment; Study Observation
Other: Questionnaire Administration — Ancillary studies
Other: Telemedicine Visit — Complete telehealth assessment visits
  Other Names: Telemedicine Encounter
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase IV trial compares patient satisfaction with telehealth versus in-person neuro-oncology assessments among glioma patients receiving oral chemotherapy. Gliomas are the most common primary central nervous system cancer and are associated with a high symptom burden, such as drowsiness, fatigue, memory difficulty, and difficulty communicating. Care at a high volume center is associated with an overall survival benefit, however, many patients may have physical or financial difficulties preventing access to these centers. Telehealth visits use computers, cameras, videoconferencing, the internet, satellite, and wireless communications to deliver healthcare, while in-person visits require the interaction to take place in the physical presence of someone else. Telehealth neuro-oncology assessments may be preferable compared to in-person assessments in glioma patients receiving oral chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess patient satisfaction with care delivered as measured by institutional Press-Ganey survey scores obtained following telehealth and in-person assessments.

SECONDARY OBJECTIVES:

I. Assess completion rate of planned oral chemotherapy among patients with glioma within 28 days of telehealth visits compared to within 28 days of in-person visits.

II. Assess preference for telehealth versus in-person neuro-oncologic evaluations among patients with glioma receiving oral chemotherapy.

III. Assess acute care utilization days, defined as emergency department evaluations and days of hospitalization within 28 days of telehealth visits compared to within 28 days of in-person visits.

IV. Assess neurologic impairment as measured by the Neurologic Assessment in Neuro-Oncology (NANO) scale will be measured at each visit with rate of neurological decline within the 28 days following telehealth assessments compared to neurological decline within the 28 days following in-person assessments.

V. Assess quality of life as measured by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30), a 30-item questionnaire that is used to assess the quality of life of cancer patients, completed at baseline and at the end of each chemotherapy cycle.

OUTLINE:

Patients receive temozolomide orally (PO) once daily (QD) on days 1-5 of each cycle. Cycles repeat every 28 days for up to 6 cycles while on study in the absence of disease progression or unacceptable toxicity. Patients complete alternating telehealth assessment visits and in-person assessment visits after each cycle of treatment.

After completion of study intervention, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of glioma requiring adjuvant chemotherapy. Patients with glioblastoma (GBM); astrocytoma, IDH-mutant; oligodendroglioma IDH-mutant, 1p/19q codeleted are eligible
* Patients eligible to receive temozolomide as standard of care adjuvant therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2, AND Karnofsky performance status (KPS) of ≥ 60
* Expected survival ≥ 6 months in the opinion of treatment team
* Willing and able to adhere with the protocol for the duration of the study including undergoing treatment, and attending scheduled visits, and examinations
* Participants who do not have devices that will permit telehealth visits will be provided such tablet devices to facilitate appointments for the duration of the study
* Participants who do not have financial resources to travel for in-person visits will be provided assistance for cost of travel
* Ability to complete patient experience surveys by the participant with or without assistance from their caregiver

Exclusion Criteria:

* Uncontrolled and/or intercurrent illness or other condition which limits safety of or compliance with study proceedings
* Pregnant or nursing, imprisoned, or lacking capacity for understanding
* Unable to swallow tablets or at risk for impaired absorption of oral medication
* Known hypersensitivity or allergy to temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with care delivered | Up to 6 months
  Satisfaction will be measured using Press-Ganey survey scores. Scores following each cycle of chemotherapy will be compared between alternating telehealth and in-person visits. The mean score associated with the telehealth visits versus (vs.) the in-person visits will be calculated for each patient. Potential patterns of changes associated with these scores over time will be graphically evaluated. Repeated measures mixed effects models will be used to further evaluate potential influence of a time element with the satisfaction scores for telehealth vs. in-person assessments.

SECONDARY OUTCOMES:
Completion rate of planned oral chemotherapy | Within 28 days of telehealth or in-person visits and up to 6 months
  The proportion of doses planned for a cycle that are completed for the telehealth vs. the in-person cycles for patients will be evaluated. The average completion rates for telehealth vs. in-person assessment cycles will be evaluated and compared across patients.
Preference for telehealth vs. in-person neuro-oncologic evaluations | Up to 6 months
  Preference will be assessed using the Visit Modality Preference Assessment, a single question with multiple choice answer (in-person visit, virtual visit, or no preference). These will be summarized both graphically and quantitatively and compared between the treatment groups.
Acute care utilization days | Within 28 days of telehealth or in-person visits, up to 6 months
  Emergency department visits and days of hospitalization compared between telehealth visits and in-person visits will be summarized both graphically and quantitatively.
Neurologic impairment - NANO | Up to 6 months
  Neurologic impairment will be measured by the Neurologic Assessment in Neuro-Oncology (NANO) scale at each visit with rate of neurological decline within the 28 days following telehealth assessments compared to neurological decline within the 28 days following in-person assessments. he NANO scale is a quick, office-based assessment that evaluates eight neurologic domains, including Gait, Strength, Upper extremity ataxia, Sensation, Visual fields, Facial strength, Language, and Level of consciousness.
Change in quality of life - EORTC QLQ-C30 | Up to 6 months
  Quality of life measures will be obtained using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) at baseline (enrollment) and following each chemotherapy cycle (28 days). The EORTC QLQ-C30 consists of three sections: functioning (15questions), symptom (13 questions), and global health status (2questions). The higher the total score, the better the quality of life; the lower the score in the symptom scale, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur T. Sener, MD, Principal Investigator — Mayo Clinic; Tufia C. Haddad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Sener U, Galloway T, Neth B, Uhm J, Kizilbash SH, Campian JL, Caron S, Breen WG, Lehrer E, Golembiewski E, Schultz S, Hughes H, Steinmetz S, Geyer S, Mead-Harvey C, Huebert C, Tauer W, Mason C, Burns TC, Pritchett J, Haddad T. Protocol for neuro-oncology anywhere 242: Pilot study evaluating telehealth and in-person assessments in patients with glioma receiving oral chemotherapy. Contemp Clin Trials Commun. 2025 Dec 23;49:101593. doi: 10.1016/j.conctc.2025.101593. eCollection 2026 Feb. PMID 41567708
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials